CLINICAL TRIAL: NCT06810336
Title: Pain Control and Quality of Recovery After Intravenous Methadone Versus Intravenous Remifentanil in Craniotomy Surgery
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Lauren Dunn, MD, Associate Professor of Anesthesiology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSR240122
Record Dates: First submitted 2025-01-23; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Brain Injury; Brain Tumors; Craniotomy Surgery; Pain; Postoperative; Postoperative Care
Keywords: craniotomy
MeSH Terms: conditions — Brain Injuries; Brain Neoplasms; Pain | interventions — Remifentanil; Methadone

STUDY DESIGN:
Intervention Model Description: a single blind study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV Remifentanil (Active Comparator): titratable medication, dosage determined by anesthesia care team.
  Interventions: Drug: Remifentanil
- IV Methadone (Experimental): 0.2 mg / kg Intravenous delivery prior to incision
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Remifentanil — Intravenous Remifentanil
  Arms: IV Remifentanil
Drug: Methadone — Intravenous Methadone
  Arms: IV Methadone

SUMMARY:
Postoperative pain is prevalent after intracranial surgery. Patients undergoing craniotomy are typically managed with short acting opioids to enable early and reliable post-operative neurological exam as well as avoid the risk of respiratory depression. However, a plethora of studies have shown that a majority of these patients experience moderate to severe pain in first 48 hours after surgery. Suboptimal pain control can lead to complications such as arterial hypertension and post-operative intracranial hemorrhage, and hence, increased morbidity and mortality.

Intravenous (IV) methadone has a long analgesic half-life and has N-methyl-D-aspartate (NMDA) receptor antagonist and serotonin and norepinephrine reuptake inhibitor (SNRI) properties. It has previously been shown to reduce postoperative opioid requirements, postoperative nausea and vomiting (PONV), and postoperative pain scores in patients that underwent orthopedic, abdominal, complex spine, and cardiac surgery. Similar findings have been shown in obstetric patients that underwent caesarean delivery under general anesthesia as well as patients that underwent gynecologic surgery and received IV methadone intraoperatively.

In a recently published retrospective study, a single intraoperative dose of IV methadone was well tolerated with lower pain scores as well as MME (oral morphine milligram equivalents) requirements for up to 72 hours after elective intracranial surgery.

IV methadone has, however, never been compared with conventional management via IV remifentanil for functional recovery in patients undergoing elective intercranial surgery.

The investigator's hypothesis is that intravenous (IV) methadone is non-inferior to IV remifentanil in patients who undergo elective intracranial surgery. It offers the advantage of being a single dose noninvasive analgesic modality that may contribute to decreasing MME consumption during the first 72 hours postoperatively, controlling postoperative pain, and improving quality of recovery after surgery.

DETAILED DESCRIPTION:
Postoperative pain is prevalent after intracranial surgery. Patients undergoing craniotomy are typically managed with short acting opioids to enable early and reliable post-operative neurological exam as well as avoid the risk of respiratory depression. However, a plethora of studies have shown that a majority of these patients experience moderate to severe pain in first 48 hours after surgery. Suboptimal pain control can lead to complications such as arterial hypertension and post-operative intracranial hemorrhage, and hence, increased morbidity and mortality.

Intravenous (IV) methadone has a long analgesic half-life and has N-methyl-D-aspartate (NMDA) receptor antagonist and serotonin and norepinephrine reuptake inhibitor (SNRI) properties. It has previously been shown to reduce postoperative opioid requirements, postoperative nausea and vomiting (PONV), and postoperative pain scores in patients that underwent orthopedic, abdominal, complex spine, and cardiac surgery. Similar findings have been shown in obstetric patients that underwent caesarean delivery under general anesthesia as well as patients that underwent gynecologic surgery and received IV methadone intraoperatively.

In a recently published retrospective study, a single intraoperative dose of IV methadone was well tolerated with lower pain scores as well as MME (oral morphine milligram equivalents) requirements for up to 72 hours after elective intracranial surgery.

IV methadone has, however, never been compared with conventional management via IV remifentanil for functional recovery in patients undergoing elective intercranial surgery.

The investigator's hypothesis is that intravenous (IV) methadone is non-inferior to IV remifentanil in patients who undergo elective intracranial surgery. It offers the advantage of being a single dose noninvasive analgesic modality that may contribute to decreasing MME consumption during the first 72 hours postoperatively, controlling postoperative pain, and improving quality of recovery after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Patients between ages 18 and 65 years old.
2. Undergoing supratentorial intracranial surgery
3. American Society of Anesthesiologists (ASA) physiological status I-III
4. Body Mass Index (BMI) between 18.5 and 45
5. Ability to understand and read English

Exclusion Criteria:

1. Being unable or unwilling to sign a consent
2. Anticipated discharge within 24 hours after surgery
3. Patients requiring Emergent Surgery
4. Preoperative usage of Methadone, or allergy to it.
5. Patients with chronic pain, requiring daily opioid use at the time of surgery, MME >60 as FDA defines opioid tolerant as 60 MME, long-acting forms of opioids such as fentanyl patch, oxycontin
6. Active or Prior Substance Use Disorder, undergoing active treatment with Medication of Opioid Use Disorder including methadone (once daily dosing), Buprenorphine (any formulation) and Naltrexone
7. Preoperative chronic renal insufficiency or failure (defined as a serum creatinine more than 2 mg/dl),
8. Pregnancy
9. Significant liver disease (cirrhosis or hepatic failure)
10. QTc >450 on preoperative electrocardiogram
11. Pulmonary disease necessitating home oxygen therapy
12. Inability to speak or read the English language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery after surgery on postoperative day 1,2,3 using QoR-15 psychometrical questionnaire (range 0-150). | 24 hours, 48 hours, 72 hours
  The Quality of Recovery-15 (QoR-15) scale is a patient-reported outcome measurement of the quality of recovery after surgery and anesthesia. The scale ranges from 0 to 150, with a higher score indicating a better quality of recovery. A score of 0 indicates extremely poor quality of recovery, while a score of 150 indicates excellent quality of recovery. The QoR-15 score can be classified into four severity classes: excellent, good, moderate, and poor recovery.

SECONDARY OUTCOMES:
Morphine Milligram Equivalent | 24 hours, 48 hours, 72 hours
  morphine milligram equivalent is a measurement of a given analgesic effect standardized to a milligram of morphine. In other words, agent X has the same effect as Y milligrams of morphine
Numeric Rating scale (NRS) pain scores (0-10) as noted over post-operative day 0, 1, 2, and 3. | 24 hours, 48 hours, 72 hours
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".
Overall Benefits of Analgesic Score (OBAS) as noted over post-operative day 0, 1, 2, and 3. | 24 hours, 48 hours, 72 hours
  The overall benefit of analgesic score (OBAS) is a daily survey that assesses a patient's satisfaction with analgesia, pain intensity, and adverse effects. To compute score, add all scores in items 1-7. Range: [0 - 28]. A low score indicates high benefit.
Complications and side effects as noted over post-operative day 0, 1, 2, and 3. | 24 hours, 48 hours, 72 hours
  Complications and side-effects:
  (a) Ability to extubate patient in the operating room (yes or no) (i) If no, Documented Time to Extubation (b) Incidence of hypoxia (requiring >2l NC O2 to maintain SpO2 > 90), respiratory depression (RR<8), and reintubation during the hospital stay after surgery (c) Time to ambulation, passing flatus, bowel movement (d) Incidence of pruritus, antiemetic medication administered - both as needed and scheduled (surrogate for PONV)
Length of Stay in Post-Anesthesia Care Unit (PACU) | 0 hours, 24 hours
Length of Stay in Hospital | From day of surgery to hospital discharge, expected to range from 5 to 10 days
  Length of stay will be recorded from the calendar day of surgery through the calendar day of hospital discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Russell T, Mitchell C, Paech MJ, Pavy T. Efficacy and safety of intraoperative intravenous methadone during general anaesthesia for caesarean delivery: a retrospective case-control study. Int J Obstet Anesth. 2013 Jan;22(1):47-51. doi: 10.1016/j.ijoa.2012.10.007. Epub 2012 Dec 7. PMID 23219678
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Marymont JH, Shear T, Parikh KN, Patel SS, Gupta DK. Intraoperative Methadone for the Prevention of Postoperative Pain: A Randomized, Double-blinded Clinical Trial in Cardiac Surgical Patients. Anesthesiology. 2015 May;122(5):1112-22. doi: 10.1097/ALN.0000000000000633. PMID 25837528
- [Background] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538
- [Background] Gourlay GK, Wilson PR, Glynn CJ. Pharmacodynamics and pharmacokinetics of methadone during the perioperative period. Anesthesiology. 1982 Dec;57(6):458-67. doi: 10.1097/00000542-198212000-00005. No abstract available. PMID 6128949
- [Background] Mancini I, Lossignol DA, Body JJ. Opioid switch to oral methadone in cancer pain. Curr Opin Oncol. 2000 Jul;12(4):308-13. doi: 10.1097/00001622-200007000-00006. PMID 10888415
- [Background] Kharasch ED. Intraoperative methadone: rediscovery, reappraisal, and reinvigoration? Anesth Analg. 2011 Jan;112(1):13-6. doi: 10.1213/ANE.0b013e3181fec9a3. No abstract available. PMID 21173206
- [Background] Basali A, Mascha EJ, Kalfas I, Schubert A. Relation between perioperative hypertension and intracranial hemorrhage after craniotomy. Anesthesiology. 2000 Jul;93(1):48-54. doi: 10.1097/00000542-200007000-00012. PMID 10861145
- [Background] Molnar L, Simon E, Nemes R, Fulesdi B, Molnar C. Postcraniotomy headache. J Anesth. 2014 Feb;28(1):102-11. doi: 10.1007/s00540-013-1671-z. Epub 2013 Jul 12. PMID 23846599
- [Background] Tsaousi GG, Logan SW, Bilotta F. Postoperative Pain Control Following Craniotomy: A Systematic Review of Recent Clinical Literature. Pain Pract. 2017 Sep;17(7):968-981. doi: 10.1111/papr.12548. Epub 2017 Feb 23. PMID 27996204
- [Background] Mordhorst C, Latz B, Kerz T, Wisser G, Schmidt A, Schneider A, Jahn-Eimermacher A, Werner C, Engelhard K. Prospective assessment of postoperative pain after craniotomy. J Neurosurg Anesthesiol. 2010 Jul;22(3):202-6. doi: 10.1097/ANA.0b013e3181df0600. PMID 20479664
- [Background] Flexman AM, Ng JL, Gelb AW. Acute and chronic pain following craniotomy. Curr Opin Anaesthesiol. 2010 Oct;23(5):551-7. doi: 10.1097/ACO.0b013e32833e15b9. PMID 20717011
- [Background] De Benedittis G, Lorenzetti A, Migliore M, Spagnoli D, Tiberio F, Villani RM. Postoperative pain in neurosurgery: a pilot study in brain surgery. Neurosurgery. 1996 Mar;38(3):466-9; discussion 469-70. doi: 10.1097/00006123-199603000-00008. PMID 8837797
- [Background] Gottschalk A, Berkow LC, Stevens RD, Mirski M, Thompson RE, White ED, Weingart JD, Long DM, Yaster M. Prospective evaluation of pain and analgesic use following major elective intracranial surgery. J Neurosurg. 2007 Feb;106(2):210-6. doi: 10.3171/jns.2007.106.2.210. PMID 17410701
- [Background] Vandse R, Vacaru A, Propp D, Graf J, Sran JK, Pillai P. Retrospective Study of the Safety and Efficacy of Intraoperative Methadone for Pain Management in Patients Undergoing Elective Intracranial Surgery. World Neurosurg. 2023 Jul;175:e969-e975. doi: 10.1016/j.wneu.2023.04.053. Epub 2023 Apr 19. PMID 37084845